CLINICAL TRIAL: NCT00494455
Title: Accuracy and Reliability of Continuous Glucose Monitoring in Critically Ill Patients With Shock Requiring Norepinephrine Therapy
Brief Title: Continuous Glucose Monitoring in Critically Ill Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Dr. Ulrike Holzinger, Medical University of Vienna
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 108/2005
Record Dates: First submitted 2007-06-27; First posted 2007-06-29 (Estimated); Last update posted 2008-02-29 (Estimated); Status verified 2007-06

CONDITIONS: Critical Illness
Keywords: critical illness; hyperglycemia; intensive insulin therapy; glucose monitoring; shock
MeSH Terms: conditions — Critical Illness; Hyperglycemia; Shock

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Continuous subcutaneous glucose monitoring in patients without shock
  Interventions: Device: continuous subcutaneous glucose monitoring
- 2 (Active Comparator): continuous subcutaneous glucose monitoring in patients with shock
  Interventions: Device: continuous subcutaneous glucose monitoring

INTERVENTIONS:
Device: continuous subcutaneous glucose monitoring — continuous subcutaneous glucose monitoring for 72h
  Other Names: CGMS (Medtronic)
  Arms: 1
Device: continuous subcutaneous glucose monitoring — continuous subcutaneous glucose monitoring for 72h
  Other Names: CGMS (Medtronic)
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether subcutaneous continuous glucose monitoring in critically ill patients is clinically feasible accurate and reliable.

DETAILED DESCRIPTION:
Hyperglycemia is is associated with more complications and higher morbidity and mortality in critically ill patients. Therefore, strict glycemic control with a target blood glucose level between 80 and 110 mg/dl is recommended. Intensive insulin therapy requires continuous intravenous insulin infusion according to an algorithm and frequent blood glucose measurements. Implementation of intensive insulin therapy increases workload for both physicians and especially for nurses.

Continuous glucose measurement would facilitate blood glucose control in critically ill patients. Numerous studies have shown accuracy of the subcutaneous continuous glucose monitoring derived glucose values compared to blood glucose measurements in diabetics. Studies evaluating the subcutaneous continuous glucose monitoring in an inpatient-population especially in an ICU-setting are rare. Therefore the aim of this study is the prospective evaluation of continuous subcutaneous glucose monitoring in critically ill patients with circulatory shock demanding norepinephrine therapy as compared to critically ill patients without shock.

ELIGIBILITY:
Inclusion Criteria:

* Admitted patients expected to stay >48h either with circulatory shock requiring norepinephrine therapy or without circulatory shock.

Exclusion Criteria:

* Admitted patients expected to stay <48h

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-04; Primary Completion 2006-04 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
correlation of continuous glucose monitoring derived glucose values and arterial blood glucose measurements in critically ill patients with and without shock | 72h

SECONDARY OUTCOMES:
influence of norepinephrine therapy, body mass index, severity of Illness (APACHE III, SAPS II) and blood glucose level on correlation | 72h

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Holzinger, MD, Principal Investigator — Medical University of Vienna, Department of Medicine III
Locations (1):
- Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Derived] Holzinger U, Warszawska J, Kitzberger R, Herkner H, Metnitz PG, Madl C. Impact of shock requiring norepinephrine on the accuracy and reliability of subcutaneous continuous glucose monitoring. Intensive Care Med. 2009 Aug;35(8):1383-9. doi: 10.1007/s00134-009-1471-y. Epub 2009 Apr 7. PMID 19350213